CLINICAL TRIAL: NCT02993120
Title: Getting to an Improved Understanding of Low-Density Lipoprotein Cholesterol and Dyslipidemia Management (GOULD) a Registry of High Cardiovascular Risk Subjects in the United States
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20150230
Record Dates: First submitted 2016-12-02; First posted 2016-12-15 (Estimated); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Medical Conditions to be Studied; Dyslipidemia; ASCVD Management
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Cohort 1: For the cohort of approximately 500 subjects taking a PCSK9i at baseline: proof consisting of a current prescription for an approved PCSK9i and subject confirmation that they have taken a PCSK9i within 30 days prior to enrollment is necessary.
- Cohort 2: • For the cohort of approximately 2000 subjects with LDL-C ≥ 100 mg/dL: confirmation of LDL-C ≥100 mg/dL with no change in LLT for 4 weeks.
- Cohort 3: For the cohort of approximately 2500 subjects with LDL-C 70-99 mg/dL: confirmation of LDL-C 70-99 mg/dL with no change in LLT for 4 weeks

SUMMARY:
This is a multicenter observational cohort study with both retrospective and prospective data collection components in subjects with ASCVD.

The purpose of this study is to better understand cholesterol treatment patterns in the context of a changing landscape in subjects with ASCVD.

DETAILED DESCRIPTION:
This is a prospective multicenter observational cohort study with retrospective component/chart review of ASCVD subjects that is designed to describe practice patterns of cholesterol management in such subjects in the US. Up to 1 year of retrospective lipid treatment, lipid measurement patterns, and CV data in subjects with ASCVD meeting inclusion/exclusion criteria at enrolled clinical sites will be captured. The retrospective data collection is being performed for the following reasons:

* Capture relevant factors related to subject's CV risk and pertinent medical history.
* Capture changes in LLT over time as related to the subject's clinical condition and medical history and adverse events to LLT Eligible subjects will be invited to enroll in chronological order of attending the clinic. The study will enroll 3 subject cohorts with the following rationale:

  1. the first cohort will consist of approximately 500 subjects on PCSK9i at the time of enrollment. The goal is to include a large enough cohort of patients receiving PCSK9i in real world clinical practice; this will allow (for the first time) to better understand the characteristics of those patients whose treatment is escalated to include PCSK9i, the therapeutic effects of PCSK9i outside of the randomized clinical trial settings, and over a prolonged duration of follow up;
  2. the second cohort will enroll approximately 2000 subjects with LDL-C levels greater than or equal to 100 mg/dL. The purpose is to include a large group of patients with established ASCVD and suboptimal LDL control in order to better understand the treatment patterns and rates of CV events in this group;
  3. the third group will enroll approximately 2500 subjects with LDL-C levels between 70 and 99 mg/dL. The purpose is to include a large group of patients with established ASCVD and more optimal control of LDL.
* To better understand patient characteristics, lipid-lowering treatment management, rates of CV events, and potential opportunities for further LLT optimization in this group. Interactive voice response system will be used to track the number of subjects in each cohort. Once a cohort is filled, no more subjects may be enrolled into it. After the first subject is enrolled and annually thereafter, physicians will fill out a questionnaire on their general use of LLT type and dose and their overall goals of lipid management. The study specific data collection points are aligned with the standard of care physician scheduled visits. Each subject will be followed through a systematic series of medical chart reviews conducted at participating clinical sites. Initial chart reviews will occur at subject enrollment with subsequent scanning of charts occurring at the site every 6 months thereafter. In addition, questionnaires will be administered to subjects every 6 months via a CATI system (wherein an interviewer will ask the subject a series of standard questions) to determine general perceptions and attitudes towards LLT. The order of questions in the questionnaire will be based on subject response. This will facilitate reports of the number of inpatient visits, outpatient visits, outpatient procedures, diagnostic tests, prescription and nonprescription medication use in the prior 6 months. Subjects will be asked to complete questionnaires even if they do not routinely see the enrolling physician or if they have switched providers.

ELIGIBILITY:
Inclusion Criteria:

Subject

* ≥ 18 years of age at signing of informed consent
* Undergoing treatment with a statin or other non-statin lipid lowering medication
* at least 1 planned visit in the next 12 months
* available for follow-up questionnaires
* established ASCVD defined as meeting at least 1 of the following criteria:

  * coronary artery disease
  * prior history of myocardial infarction
  * coronary or other arterial revascularization
  * ischemic stroke or transient ischemic attack
  * documented peripheral arterial disease secondary to atherosclerosis (eg., aortic aneurysm, ankle brachial index < 0.9, imaging evidence of > 50% stenosis in any peripheral artery, or intermittent claudication)
  * carotid artery stenosis
  * LDL-C levels>69 mg/dL except in subjects assigned to the PCSK9i cohort Cohorts
* Cohorts are assigned based upon most recent LDL-C level prior to enrollment
* For the cohort of approximately 500 subjects taking a PCSK9i at baseline: proof consisting of a current prescription for an approved PCSK9i and subject confirmation that they have taken a PCSK9i within 30 days prior to enrollment is necessary
* For the cohort of approximately 2000 subjects with LDL-C ≥ 100 mg/dL: confirmation of LDL-C ≥ 100 mg/dL with no change in LLT for 4 weeks.
* For the cohort of approximately 2500 subjects with LDL-C 70-99 mg/dL: confirmation of LDL-C 70-99 mg/dL with no change in LLT for 4 weeks.

Exclusion Criteria:

Subject

* Unable or unwilling to provide informed consent including but not limited to cognitive or language barriers
* Current or planned participation in an interventional clinical study involving any investigational medical device or drug treatment at the time of enrollment or in the 6 months prior to enrollment. Subjects who chose to participate in an interventional clinical study of either device or drug treatment after enrollment will be removed from the GOULD study
* Life expectancy < 12 months
* Currently pregnant, breast feeding, or planning to become pregnant

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Adults (18-44 years)
  * Adults (45-64 years)
  * Adults (65-74 years)
  * Adults (75 years and older)
  * Sex: Male and Female
Sampling Method: Probability Sample
Enrollment: 5006 (Actual)
Dates: Start 2016-12-06 (Actual); Primary Completion 2021-08-06 (Actual); Study Completion 2021-08-06 (Actual)

PRIMARY OUTCOMES:
Low-density lipoprotein (LDL) treatment patterns | Through study completion, an average of 3 years
  Describe low-density lipoprotein (LDL) treatment patterns over time in subjects with clinical ASCVD

SECONDARY OUTCOMES:
LDL-C levels and measurement patterns | Through study completion, an average of 3 years
  Describe LDL-C levels and measurement patterns in subjects with clinical ASCVD
Subject Characteristics | Through study completion, an average of 3 years
  Describe subject characteristics
Subject understanding of CV risk | Through study completion, an average of 3 years
  Describe subject understanding of CV risk
Goals of Lipid Management | Through study completion, an average of 3 years
  Describe subject goals of lipid management
Attitudes towards lipid lowering treatment (LLT) | Through study completion, an average of 3 years
  Describe subject attitudes towards lipid lowering treatment (LLT)
Percentage of Subjects Achieving Pre-Specified Levels Low-Density Lipoprotein Cholesterol (LDL-C) Before and After Educational Intervention | Up to 1 Year
  The two levels of LDL-C that will be assessed are < 70 mg/dL and < 55 mg/dL.
Number of Subjects who Experience an Intensification in Lipid-Lowering Therapy Before and After Educational Intervention | Up to 1 Year
Percentage of Subjects on Optimal Medical Therapy Before and After Educational Intervention | Up to 1 Year
Percentage of Physicians Stating a Specific Lipid Treatment Objective Before and After Educational Intervention | Up to 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (104):
- United States (104):
  - Research Site, Chandler, Arizona
  - Research Site, Glendale, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Canoga Park, California
  - Research Site, Cerritos, California
  - Research Site, Los Angeles, California
  - Research Site, Oxnard, California
  - Research Site, Rancho Mirage, California
  - Research Site, Sacramento, California
  - Research Site, Wildomar, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Lafayette, Colorado
  - Research Site, Bloomfield, Connecticut
  - Research Site, Bridgeport, Connecticut
  - Research Site, Hartford, Connecticut
  - Research Site, Stamford, Connecticut
  - Research Site, Boca Raton, Florida
  - Research Site, Brandon, Florida
  - Research Site, Brooksville, Florida
  - Research Site, Daytona Beach, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Homestead, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Jacksonville Beach, Florida
  - Research Site, Miami, Florida
  - Research Site, Miami Beach, Florida
  - Research Site, Naples, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Pensacola, Florida
  - Research Site, Rockledge, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Cumming, Georgia
  - Research Site, Smyrna, Georgia
  - Research Site, Boise, Idaho
  - Research Site, Coeur d'Alene, Idaho
  - Research Site, Meridian, Idaho
  - Research Site, Nampa, Idaho
  - Research Site, Arlington Heights, Illinois
  - Research Site, Chicago, Illinois
  - Research Site, Evanston, Illinois
  - Research Site, Morton, Illinois
  - Research Site, Evansville, Indiana
  - Research Site, Michigan City, Indiana
  - Research Site, Davenport, Iowa
  - Research Site, Des Moines, Iowa
  - Research Site, Covington, Kentucky
  - Research Site, Alexandria, Louisiana
  - Research Site, Eunice, Louisiana
  - Research Site, Monroe, Louisiana
  - Research Site, Portland, Maine
  - Research Site, Baltimore, Maryland
  - Research Site, Elkridge, Maryland
  - Research Site, Great Barrington, Massachusetts
  - Research Site, Natick, Massachusetts
  - Research Site, Worcester, Massachusetts
  - Research Site, Alpena, Michigan
  - Research Site, Detroit, Michigan
  - Research Site, Flint, Michigan
  - Research Site, Grand Rapids, Michigan
  - Research Site, Lansing, Michigan
  - Research Site, Coon Rapids, Minnesota
  - Research Site, Minneapolis, Minnesota
  - Research Site, Port Gibson, Mississippi
  - Research Site, Columbia, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Lincoln, Nebraska
  - Research Site, Omaha, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Cedar Knolls, New Jersey
  - Research Site, Albany, New York
  - Research Site, Buffalo, New York
  - Research Site, Kingston, New York
  - Research Site, Rochester, New York
  - Research Site, Greensboro, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Fargo, North Dakota
  - Research Site, Columbus, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Downingtown, Pennsylvania
  - Research Site, Doylestown, Pennsylvania
  - Research Site, Jersey Shore, Pennsylvania
  - Research Site, Levittown, Pennsylvania
  - Research Site, Wynnewood, Pennsylvania
  - Research Site, Providence, Rhode Island
  - Research Site, Charleston, South Carolina
  - Research Site, Greer, South Carolina
  - Research Site, Murrells Inlet, South Carolina
  - Research Site, Summerville, South Carolina
  - Research Site, Oak Ridge, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Humble, Texas
  - Research Site, Kingwood, Texas
  - Research Site, Lufkin, Texas
  - Research Site, McKinney, Texas
  - Research Site, Mesquite, Texas
  - Research Site, Missouri City, Texas
  - Research Site, Sugar Land, Texas
  - Research Site, Tomball, Texas
  - Research Site, Hopewell, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Winchester, Virginia
  - Research Site, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Arnold SV, de Lemos JA, Rosenson RS, Ballantyne CM, Liu Y, Mues KE, Alam S, Elliott-Davey M, Bhatt DL, Cannon CP, Kosiborod M; GOULD Investigators. Use of Guideline-Recommended Risk Reduction Strategies Among Patients With Diabetes and Atherosclerotic Cardiovascular Disease. Circulation. 2019 Aug 13;140(7):618-620. doi: 10.1161/CIRCULATIONAHA.119.041730. Epub 2019 Jun 7. No abstract available. PMID 31174429
- [Background] Arnold SV, Cannon CP, de Lemos JA, Rosenson RS, Ballantyne CM, Liu Y, Alam S, Mues KE, Bhatt DL, Kosiborod M; GOULD Investigators. What Do US Physicians and Patients Think About Lipid-Lowering Therapy and Goals of Treatment? Results From the GOULD Registry. J Am Heart Assoc. 2021 Aug 17;10(16):e020893. doi: 10.1161/JAHA.120.020893. Epub 2021 Aug 7. PMID 34369165
- [Background] Cannon CP, de Lemos JA, Rosenson RS, Ballantyne CM, Liu Y, Yazdi D, Elliott-Davey M, Mues KE, Bhatt DL, Kosiborod MN; GOULD Investigators. Getting to an ImprOved Understanding of Low-Density Lipoprotein-Cholesterol and Dyslipidemia Management (GOULD): Methods and baseline data of a registry of high cardiovascular risk patients in the United States. Am Heart J. 2020 Jan;219:70-77. doi: 10.1016/j.ahj.2019.10.014. Epub 2019 Oct 31. PMID 31726422
- [Background] Arnold SV, de Lemos JA, Liu Y, Mues KE, Bhatt DL, Cannon CP, Kosiborod M. Adherence to Guideline Medication Recommendations to Prevent Atherosclerotic Cardiovascular Disease Progression Among Adults With Prior Myocardial Infarction. JAMA Netw Open. 2020 Apr 1;3(4):e203032. doi: 10.1001/jamanetworkopen.2020.3032. PMID 32301989
- [Background] Shaik A, Kosiborod M, de Lemos JA, Gao Q, Mues KE, Alam S, Bhatt DL, Cannon CP, Ballantyne CM, Rosenson RS; GOULD Investigators. Use of lipid-lowering therapies in patients with chronic kidney disease and atherosclerotic cardiovascular disease: 2-year results from Getting to an imprOved Understanding of Low-Density lipoprotein cholesterol and dyslipidemia management (GOULD). Clin Cardiol. 2022 Dec;45(12):1303-1310. doi: 10.1002/clc.23923. Epub 2022 Sep 19. PMID 36124341
- [Background] Arnold SV, de Lemos JA, Zheng L, Rosenson RS, Ballantyne CM, Alam S, Bhatt DL, Cannon CP, Kosiborod M; GOULD Investigators. Use of optimal medical therapy in patients with diabetes and atherosclerotic cardiovascular disease: Insights from a prospective longitudinal cohort study. Diabetes Obes Metab. 2023 Jun;25(6):1750-1757. doi: 10.1111/dom.15032. Epub 2023 Mar 7. PMID 36843558
- [Background] Peterson BE, Bhatt DL, Ballantyne CM, de Lemos JA, Rosenson RS, Kosiborod MN, Cannon CP; GOULD Investigators. Intensity of Lipid-Lowering Therapy Among Patients With Polyvascular Disease. JAMA Netw Open. 2023 Mar 1;6(3):e234709. doi: 10.1001/jamanetworkopen.2023.4709. PMID 36972054
- [Derived] Cannon CP, Ballantyne CM, Bhatt DL, de Lemos JA, Gao Q, Kui N, Rosenson RS, Mues KE, Exter J, Alam S, Kosiborod MN; GOULD EDU Investigators. GOULD EDU: Cluster-Randomized Trial of an Educational Intervention to Improve Lipid-Lowering Guideline Adherence. JACC Adv. 2026 Jan;5(1):102403. doi: 10.1016/j.jacadv.2025.102403. Epub 2025 Dec 3. PMID 41344145
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com